CLINICAL TRIAL: NCT01602510
Title: A Fixed-Dose Study of Lamotrigine Versus Placebo in the Long Term Prevention of Relapse and/or Recurrence of a Manic, Hypomanic, Mixed or Depressive Episode in Adult Subjects With Bipolar I Disorder
Brief Title: Lamotrigine Phase III Study in Bipolar I Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 113783
Record Dates: First submitted 2012-05-17; First posted 2012-05-21 (Estimated); Results first posted 2017-01-23 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2016-09

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Lamotrigine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Lamotrigine CD (Experimental): lamotrigine chewable dispersible tablets 25mg, 50mg, 100mg
  Interventions: Drug: Lamotrigine
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lamotrigine — in the double blind phase, lamotrigine 200mg/day will be used among half of eligible subjects after randomization
  Arms: Lamotrigine CD
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This registration study in China is a multi-centre, double-blind, placebo-controlled clinical trial to evaluate the efficacy and safety of lamotrigine in the prevention of recurrence/relapse of mood episodes in subjects with bipolar I disorder. Subjects are bipolar I disorder patients with recent/current manic, hypomanic, mixed or depressive episode. The study will include an open-label phase and a randomized phase. During the open-label phase, subjects will have lamotrigine monotherapy or combination therapy escalation. The target dose of lamotrigine is 200 milligram (mg)/day monotherapy. The duration of treatment in the open-label phase will last 6-16 weeks, until subjects reach a stable dose of lamotrigine. Beginning at week 7 of the open-label phase, subjects who have reached a stable dose of lamotrigine and met response criteria, defined as maintaining a Clinical Global Impression of Severity (CGI-S) score <= 3 for at least 4 continuous weeks and maintaining lamotrigine 200 mg/day monotherapy for at least 1 week, will be eligible to enroll in the double-blind phase of the study. Subjects who have not met response criteria after 16 weeks of participation in the open-label phase will be withdrawn from the study. Subjects will have lamotrigine 200 mg/day monotherapy for at least 1 week prior to randomization. Subjects who have met randomization requirements will be randomized 1:1 to lamotrigine 200 mg/day or placebo for 36 weeks double-blind treatment. After randomization, subjects will be assessed at weekly intervals for the first month, biweekly intervals for the second month, and then at monthly intervals for up to 36 weeks of double-blind treatment. The primary endpoint will be TIME, defined as the time to intervention (addition of pharmacotherapy or electroconvulsive therapy [ECT]) for any mood episode (relapse or recurrence of a depressive, manic, hypomanic or mixed episode) after randomization. The secondary endpoints will include time to intervention for manic, hypomanic or mixed episode (TIMan) and time to intervention for depressive episode (TIDep).The scores on the Hamilton Depression (HAMD), Young Mania Rating Scale (YMRS), CGI-I, CGI-S and Global Assessment Scale (GAS) will be used as indicators for both intensity and duration of mood symptoms during this phase. Subjects who withdraw early from the study prior to week 36 or reach TIME will have a follow-up visit 14 days after the last dose of investigational drug.

ELIGIBILITY:
Inclusion Criteria:

For open label phase

* Subjects must be able to effectively communicate with study personnel, have the ability to comprehend the key components of the Inform Consent Form and must provide written informed consent to participate in the study prior to any study-specific assessments or procedures.
* An in-patient or out-patient (male or female) and aged >=18 years old.
* Disease to be studied: Has a diagnosis of the following disease as defined by DSM-IV criteria currently or within 60 days:

  a)Bipolar I Disorder, most recent episode depressed (296.5x); b)Bipolar I Disorder, most recent episode hypomanic (296.40); c)Bipolar I Disorder, most recent episode manic (296.4x); d)Bipolar I Disorder, most recent episode mixed (296.6x)
* The subject who has a diagnose of "bipolar I disorder, most recent episode depressed (296.5x)" must meet the following criteria:

Has at least one well documented manic, hypomanic or mixed episode, as defined by DSM-IV criteria, within 3 years of enrolment ; The duration of recent/current depressive episode is at least 2 weeks but not longer than 12 months prior to enrolment; For subject with currently experiencing a depressive episode, he/she must have a minimum total score of 18 on the HAMD-17 at s screening.

- The subject who has a diagnosis of "bipolar I disorder, most recent episode hypomanic (296.40)" or "bipolar I disorder, most recent episode manic (296.4x)" or "bipolar I disorder, most recent episode mixed (296.6x)" must meet the following criteria: Has had at least one well documented additional manic, hypomanic or mixed episode and one depressed episode, as defined by DSM-IV criteria, within 3 years of enrolment; Has a duration of the index manic episode of at least 1 week (unless hospitalised) or hypomanic episode of at least 4 days or mixed episode of at least 1 week. In neither case should the index episode be more than 12 months in duration; If the subject's index episode is the subject's initial/current manic mood event, subject must have a minimum score of 10 on the first 11 items of the YMRS at screening; If the subject's index episode is the subject's initial/current mixed mood event, subject must have a minimum score of 10 on the first 11 items of the YMRS, and have a minimum score of 18 on the HAMD-17 at screening.

For randomized double-blind phase

* Has been on Lamotrigine 200 mg/day monotherapy for at least 1 week.
* CGI-S score <= 3 for at least 4 continuous weeks of treatment prior to randomization.
* Has demonstrated adequate compliance with IP (compliance rate: 75%-125%, inclusive).

Exclusion Criteria:

For open label

* Has met Diagnostic and Statistical Manual of Mental Disorders-IV (DSM-IV) criteria for rapid cycling and has had more than 4 manic, hypomanic, mixed or depressive episodes in the 12-month period prior to enrollment.
* Has a significant DSM-IV Axis II diagnosis which would suggest non-responsiveness to pharmacotherapy for bipolar disorder or non-compliance with the protocol.
* Has a current or previous diagnosis of an Axis I disorder (including anorexia nervosa or bulimia nervosa) with the exception of bipolar disorder or has received corresponding treatment, or has been diagnosed with dysthymia within the previous 2 years.
* Has signs or symptoms of psychosis.
* The subject, in the investigator's judgment, poses a suicidal risk, has attempted suicide within 6 months prior to screening (assessed using the Columbia Suicide Severity Rating Scale Baseline) or .
* Has documented Intelligence quotient < 70 or suspected mental retardation.
* Has a history of substance abuse or dependence within 12 months prior to enrolment (DSM-IV defined substance categories, excluding nicotine and caffeine and including alcohol), or has as a positive urine test for illicit drug use (excluding nicotine and caffeine).
* Has received fluoxetine within 4 weeks prior to entry into the open-label phase; has received oral contraceptives or other hormonal preparations containing estrogen within 2 weeks prior to entry into the open-label phase; has received lopinavir/ritonavir or atazanavir /ritonavir within 7 days prior to the baseline visit.
* Has a clinically significant and/or unstable medical disorder (with or without lab test results); or clinically significant test results (thyroid function, electrocardiogram, hematology, clinical chemistry, or urinalysis) as per investigator's judgment; or a disorder that would interfere with the action, absorption, distribution, metabolism, or excretion of lamotrigine; per investigator's clinical judgment (after consulting GSK medical monitor), might pose a safety concern; or interfere with the accurate assessment of safety or efficacy.
* Has a history or current diagnosis of epilepsy.
* Is morbidly obese, i.e. if Body Mass Index (BMI) is > 35 {BMI = Body weight (in kg) divided by (Height in meters squared).
* Single or average QT interval corrected by Bazette's formulaQTcB or QTc > 450 millisecond (msec); for patients with bundle branch block QTc > 480 msec.
* Has a history of hepatic dysfunction; Alanine aminotransferase (ALT) or Aspartate aminotransferase (AST) >= 2 x upper limit of normal (ULN); Alkaline phosphatase (ALP) or total bilirubin > 1.5 x ULN (excluding total bilirubin > 1.5 x ULN but direct bilirubin < 35%) or other conditions which, in the investigator's judgment, would render patients unsuitable for the study.
* Has a history of drug allergy (including rash) or a medically significant adverse effect from any ingredient of lamotrigine, or a history of rash due to anti-epileptic drugs or has frequent and/or serious hypersensitivity reaction to multiple drugs.
* Participation in any study related to lamotrigine within 6 months before screening or has received lamotrigine within 4 weeks before screening.
* Participation in another clinical study unrelated to the current illness currently or within the previous 30 days, or 3 months for studies related to the current illness.
* Initiation of systematic psychotherapy within 3 months prior to screening or planned initiation of systematic psychotherapy during the study.
* Female subjects who are pregnant, lactating or do not agree to use the contraceptive methods such as use of condom, injection of progesterone, a reliable barrier method of birth control, partner with vasectomy or abstinence during the study.

For randomized double blind phase

* Has signs or symptoms of psychosis.
* Requires treatment for a manic or mixed episode in the open-label phase with new courses of lithium, psychotropic drugs or other drugs with a half-life greater than 14 days.
* Has become actively suicidal and/or has a score >=3 on item 3 of the HAMD.
* Has tested positive for an illicit drug on lab analysis administered before randomization or alcohol abuse/addiction.
* Has had a change in lamotrigine dosage during the last week of the open-label phase.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2012-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (16):
- China (16):
  - GSK Investigational Site, Guangzhou, Guangdong
  - GSK Investigational Site, Baoding, Hebei
  - GSK Investigational Site, Shijiazhuang, Hebei
  - GSK Investigational Site, Harbin, Heilongjiang
  - GSK Investigational Site, Changshacun, Henan
  - GSK Investigational Site, Xinxiang, Henan
  - GSK Investigational Site, Wuhan, Hubei
  - GSK Investigational Site, Changsha, Hunan
  - GSK Investigational Site, Nanjing, Jiangsu
  - GSK Investigational Site, Xi'an, Shaanxi
  - GSK Investigational Site, Taiyuan, Shanxi
  - GSK Investigational Site, Chengdu, Sichuan
  - GSK Investigational Site, Kunming, Yunnan
  - GSK Investigational Site, Hangzhou, Zhejiang
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Shanghai

REFERENCES:
- [Derived] Zhang L, Zhang H, Lv LX, Tan Q, Xu X, Hu J, Zi L, Cooper J, Phansalkar A, Wang G. A randomised, double-blind, placebo-controlled study to evaluate the safety and efficacy of lamotrigine in the maintenance treatment of Chinese adult patients with bipolar I disorder. Int J Bipolar Disord. 2022 Aug 1;10(1):20. doi: 10.1186/s40345-022-00266-4. PMID 35909213

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study consisted of 4 phases: screen phase (<2 weeks[W]), open-label phase (OLP) (Up to 16 W, lamotrigine monotherapy (LM) or combination therapy escalated to a target dose of LM 200 milligrams [mg]/day[D]), randomized double-blind phase (RDP) (up to 36 W, lamotrigine 200 mg/day or placebo) and follow-up visit (14 days after the last dose).
Pre-assignment Details: 420 participants entered into OLP and received at least one dose of study medication. Of these 420 participants, 264 were randomized into RDP.
Groups:
- Open Label Lamotrigine 200 mg/Day: Participants (Par.) received lamotrigine escalated to a target dose of lamotrigine 200mg/day monotherapy for 6 weeks to 16 weeks. If needed, concomitant psychotropic medications were permitted during this phase however medications were discontinued at least 1 week before entering into the double-blind phase.
- Randomized Placebo: Participants who reached a stable dose of lamotrigine and met response criteria, defined as a Clinical Global Impression of Severity (CGI-S) score <= 3 maintained for at least 4 continuous weeks and lamotrigine 200 mg/day monotherapy maintained for at least 1 week during open label phase, were enrolled in the double-blind phase of the study. Participants received placebo for 36 weeks.
- Randomized Lamotrigine 200 mg/Day: Participants who reached a stable dose of lamotrigine and met response criteria, defined as a CGI-S score <= 3 maintained for at least 4 continuous weeks and lamotrigine 200 mg/day monotherapy maintained for at least 1 week during open label phase, were enrolled in the double-blind phase of the study. Participants received lamotrigine 200 mg/day for 36 weeks.
Period: Open Label Phase
Arm/Group | Open Label Lamotrigine 200 mg/Day | Randomized Placebo | Randomized Lamotrigine 200 mg/Day
Started | 420 | 0 | 0
Completed | 117 | 0 | 0
Not Completed | 303 | 0 | 0
Not completed — Adverse Event | 46 | 0 | 0
Not completed — Lack of Efficacy | 22 | 0 | 0
Not completed — Protocol Violation | 15 | 0 | 0
Not completed — Met protocol-defined stopping criteria | 122 | 0 | 0
Not completed — Lost to Follow-up | 22 | 0 | 0
Not completed — Physician Decision | 19 | 0 | 0
Not completed — Withdrawal by Subject | 57 | 0 | 0
Period: Randomized Phase
Arm/Group | Open Label Lamotrigine 200 mg/Day | Randomized Placebo | Randomized Lamotrigine 200 mg/Day
Started | 0 | 133 | 131
Completed | 0 | 59 | 58
Not Completed | 0 | 74 | 73
Not completed — Adverse Event | 0 | 2 | 6
Not completed — Lack of Efficacy | 0 | 4 | 4
Not completed — Protocol Violation | 0 | 3 | 3
Not completed — Met protocol-defined stopping criteria | 0 | 58 | 48
Not completed — Lost to Follow-up | 0 | 1 | 3
Not completed — Physician Decision | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 6 | 7

BASELINE CHARACTERISTICS:
Groups:
- Open Label Lamotrigine 200 mg/Day: Participants (Par.) received lamotrigine escalated to a target dose of lamotrigine 200 mg/day monotherapy for 6 weeks to 16 weeks. If needed, concomitant psychotropic medications were permitted during this phase however medications were discontinued at least 1 week before entering into the double-blind phase.
Arm/Group | Open Label Lamotrigine 200 mg/Day
Number analyzed (Participants) | 420
Age, Continuous [Mean (Standard Deviation); unit: Years] — Data is presented for Open Label Phase.
  Years | 35.7 (11.72)
Gender [Count of Participants; unit: Participants] — Data is presented for Open Label Phase.
  Participants
    Female | 220
    Male | 200
Race/Ethnicity, Customized [Number; unit: Participants] — Data is presented for Open Label Phase.
  Participants
    Not Hispanic or Latino | 420

OUTCOME MEASURES:

1. Primary Outcome: Time to Intervention for Any Mood Episode (TIME)
Description: TIME is defined as being the time from entry into the randomized double-blind phase to the time of the first prescription of any additional pharmacotherapy or Electroconvulsive therapy (ECT) determined by the investigator to be necessary for treatment of a relapse and/or recurrence of a depressive, manic, hypomanic or mixed episode, whichever occurs first. TIME was measured relative to randomization date. Par. prematurely discontinued from the study prior to reaching the TIME event were censored at the time of discontinuation. Analysis was performed using Cox proportional hazards regression model with covariates of site, CGI-S baseline score, treatment and treatment by CGI-S baseline score interaction. The overall hazard ratio for treatment group could not be calculated due to different CGI-S baseline score level.
Time Frame: 36 weeks (wks)
Population: Randomized (RD) Full analysis population: comprised of all randomized par. who took at least one dose of study medication and had at least one post-baseline efficacy/health outcomes assessment during randomized double-blind phase. "NA" implies no data are available. Only those par. with available data at indicated time points were analyzed.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Randomized Placebo | Randomized Lamotrigine 200 mg/Day
Number analyzed (Participants) | 62 | 50
Days | NA [NA to NA] — With less than 50% of the Participants got TIME events the median and corresponding 95% confidence interval can not be calculated | NA [NA to NA] — With less than 50% of the Participants got TIME events the median and corresponding 95% confidence interval can not be calculated
Statistical Analysis 1: Comparison: Randomized Placebo vs Randomized Lamotrigine 200 mg/Day; Test type: Superiority or Other; p = 0.438, Regression, Cox; Adjusted Hazard Ratio = 0.86, 95% CI 2-sided [0.59 to 1.25] — p value with Treatment Group as covariate
Statistical Analysis 2: Comparison: Randomized Placebo vs Randomized Lamotrigine 200 mg/Day; Test type: Superiority or Other; p = 0.212, Regression, Cox; Adjusted Hazard Ratio = 0.86, 95% CI 2-sided [0.59 to 1.25] — p value with Site as covariate
Statistical Analysis 3: Comparison: Randomized Placebo vs Randomized Lamotrigine 200 mg/Day; Test type: Superiority or Other; p = 0.724, Regression, Cox; Adjusted Hazard Ratio = 0.86, 95% CI 2-sided [0.59 to 1.25] — p value with CGI-S Baseline Score as covariate

2. Secondary Outcome: Time to Intervention for Manic, Hypomanic or Mixed Episode (TIMan)
Description: TIMan was analyzed using using Cox proportional hazards regression model with covariates of site, CGI-S baseline score, treatment and treatment by CGI-S baseline score interaction. The overall hazard ratio for treatment group could not be calculated due to different CGI-S baseline score level. Par. prematurely discontinued from the study prior to reaching the event were censored at the time of discontinuation.
Time Frame: 36 weeks
Population: RD Full Analysis Population."NA" implies no data are available. Only those par. with available data at indicated time points were analyzed.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Randomized Placebo | Randomized Lamotrigine 200 mg/Day
Number analyzed (Participants) | 27 | 24
Days | NA [NA to NA] — With less than 50% of the Participants got TIMan events the median and corresponding 95% confidence interval can not be calculated | NA [NA to NA] — With less than 50% of the Participants got TIMan events the median and corresponding 95% confidence interval can not be calculated
Statistical Analysis 1: Comparison: Randomized Placebo vs Randomized Lamotrigine 200 mg/Day; Test type: Superiority or Other; p = 0.869, Regression, Cox; Adjusted Hazard Ratio = 0.95, 95% CI 2-sided [0.55 to 1.66] — p value with Treatment Group as covariate
Statistical Analysis 2: Comparison: Randomized Placebo vs Randomized Lamotrigine 200 mg/Day; Test type: Superiority or Other; p = 0.061, Regression, Cox; Adjusted Hazard Ratio = 0.95, 95% CI 2-sided [0.55 to 1.66] — p value with Site as covariate
Statistical Analysis 3: Comparison: Randomized Placebo vs Randomized Lamotrigine 200 mg/Day; Test type: Superiority or Other; p = 0.505, Regression, Cox; Adjusted Hazard Ratio = 0.95, 95% CI 2-sided [0.55 to 1.66] — p value with CGI-S Baseline Score as covariate

3. Secondary Outcome: Time to Intervention for Depressive Episode (TIDep)
Description: TIDep was analyzed using Cox proportional hazards regression model with covariates of site, CGI-S baseline score, treatment and treatment by CGI-S baseline score interaction. The overall hazard ratio for treatment group could not be calculated due to different CGI-S baseline score level. Par. prematurely discontinued from the study prior to reaching the event were censored at the time of discontinuation.
Time Frame: 36 weeks
Population: RD Full Analysis Population. "NA" implies no data are available. Only those par. with available data at indicated time points were analyzed.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Randomized Placebo | Randomized Lamotrigine 200 mg/Day
Number analyzed (Participants) | 35 | 26
Days | NA [NA to NA] — With less than 50% of the Participants got TIDep events the median and corresponding 95% confidence interval can not be calculated | NA [NA to NA] — With less than 50% of the Participants got TIDep events the median and corresponding 95% confidence interval can not be calculated
Statistical Analysis 1: Comparison: Randomized Placebo vs Randomized Lamotrigine 200 mg/Day; Test type: Superiority or Other; p = 0.369, Regression, Cox; Adjusted Hazard Ratio = 0.79, 95% CI 2-sided [0.48 to 1.32] — p value with Treatment Group as covariate
Statistical Analysis 2: Comparison: Randomized Placebo vs Randomized Lamotrigine 200 mg/Day; Test type: Superiority or Other; p = 0.955, Regression, Cox; Adjusted Hazard Ratio = 0.79, 95% CI 2-sided [0.48 to 1.32] — p value with Site as covariate
Statistical Analysis 3: Comparison: Randomized Placebo vs Randomized Lamotrigine 200 mg/Day; Test type: Superiority or Other; p = 0.874, Regression, Cox; Adjusted Hazard Ratio = 0.79, 95% CI 2-sided [0.48 to 1.32] — p value with CGI-S Baseline Score as covariate

4. Secondary Outcome: Overall Survival in Study (TIME-SIS).
Description: TIME-SIS was defined as the time to intervention (addition of pharmacotherapy or ECT) for any mood episode, or to the time when the participant is withdrawn for any reason after randomization. The premature discontinuation of a participant prior to reaching TIME, for any reason, was treated as an event related to bipolar disorder. All participants prematurely discontinued prior to the TIME event in this analysis were to be assumed to have reached TIME. TIMS-SIS was analyzed using Cox proportional hazards regression model with covariates of site, CGI-S baseline score, treatment and treatment by CGI-S baseline score interaction. The overall hazard ratio for treatment group could not be calculated due to different CGI-S baseline score level. Par. prematurely discontinued from the study prior to reaching the event were censored at the time of discontinuation.
Time Frame: 36 weeks
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Randomized Placebo | Randomized Lamotrigine 200 mg/Day
Number analyzed (Participants) | 75 | 72
Days | 183 [140 to NA] — With less than 50% of the Participants got TIME events the upper bound of 95% confidence interval for median can not be calculated. | 188 [117 to NA] — With less than 50% of the Participants got TIME events the upper bound of 95% confidence interval for median can not be calculated.
Statistical Analysis 1: Comparison: Randomized Placebo vs Randomized Lamotrigine 200 mg/Day; Test type: Superiority or Other; p = 0.927, Regression, Cox; Adjusted Hazard Ratio = 1.02, 95% CI 2-sided [0.73 to 1.40] — p value with Treatment Group as covariate
Statistical Analysis 2: Comparison: Randomized Placebo vs Randomized Lamotrigine 200 mg/Day; Test type: Superiority or Other; p = 0.036, Regression, Cox; Adjusted Hazard Ratio = 1.02, 95% CI 2-sided [0.73 to 1.40] — p value with Site as covariate
Statistical Analysis 3: Comparison: Randomized Placebo vs Randomized Lamotrigine 200 mg/Day; Test type: Superiority or Other; p = 0.509, Regression, Cox; Adjusted Hazard Ratio = 1.02, 95% CI 2-sided [0.73 to 1.40] — p value with CGI-S Baseline Score as covariate

5. Secondary Outcome: Change From Baseline in Clinical Global Impression of Improvements (CGI-I)
Description: The CGI-I is a 7-point scale where investigator were asked to assess the participant's illness at the time of assessment (improved or worsened) relative to a baseline state. In this scale, 1= very much improved; 2= much improved; 3= minimally improved; 4= no change; 5= minimally worse; 6= much worse; or 7= very much worse. Analysis was performed using Analysis of covariance with covariates of site, CGI-S baseline score and treatment. In presented Last-observation-carried-forward datasets, the last non-missing on therapy (OT) score prior to TIME was carried forward to estimate missing data points for the remaining study visits of the treatment period. Baseline value was defined as the last non-missing values at or prior to the randomization. Change from baseline at the time point of interest was calculated by subtracting the baseline values from the individual post-baseline values. If either baseline or post-baseline value was missing, the change from baseline was set to missing.
Time Frame: Baseline and up to 36 weeks
Population: RD Full Analysis Population.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Randomized Placebo | Randomized Lamotrigine 200 mg/Day
Number analyzed (Participants) | 133 | 130
Score on a scale | 2.6 (0.20) | 2.7 (0.21)
Statistical Analysis 1: Comparison: Randomized Placebo vs Randomized Lamotrigine 200 mg/Day; Test type: Superiority or Other; p = 0.833, ANCOVA; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.4 to 0.5]

6. Secondary Outcome: Change From Baseline in Clinical Global Impression of Severity (CGI-S)
Description: The CGI-S is a 7-point scale where investigator were asked to rate the severity of the participant's illness at the time of assessment on severity of mental illness, where 1= normal, and 7= extremely ill. Data was collected on Weeks 0, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 32 and 36. Analysis performed using Analysis of Covariance (ANCOVA) with covariates of site, CGI-S baseline score (Open label phase), treatment and CGI-S baseline score. In presented Last observation carried forward (LOCF) datasets, last non-missing on therapy score prior to TIME was carried forward to estimate missing data points for remaining study visits of treatment period. The baseline value was defined as last non-missing values at or prior to the randomization. The change from baseline at the time point of interest was calculated by subtracting the baseline values from individual post-baseline values. If either the baseline or post-baseline value was missing, the change from baseline was set to missing as well.
Time Frame: Baseline and up to 36 weeks
Population: RD Full Analysis Population.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Randomized Placebo | Randomized Lamotrigine 200 mg/Day
Number analyzed (Participants) | 133 | 130
Score on a scale | 0.7 (0.15) | 0.5 (0.15)
Statistical Analysis 1: Comparison: Randomized Placebo vs Randomized Lamotrigine 200 mg/Day; Test type: Superiority or Other; p = 0.245, ANCOVA; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.5 to 0.1]

7. Secondary Outcome: Change From Baseline in Hamilton Depression Rating Scale (HAMD)
Description: HAMD consists of 17 items: depressed mood, feelings of guilt, suicide, insomnia-early, middle, late, work and activities, retardation, agitation, anxiety psychic, anxiety somatic, somatic symptoms gastro-intestinal, general somatic symptoms, hypochondriasis, loss of weight, and insight. Investigators rated par. from 0 to 4 (or 2) for these items. Total score is sum of all subscales (0 to 52, higher is worse). Data was collected on Wks 0, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 32, 36. Analysis was performed using ANCOVA with covariates of site, CGI-S baseline (BL) score, treatment and HAMD total BL score. The last non-missing OT score prior to TIME was carried forward to estimate missing data points for remaining study visits of the treatment period. BL value was defined as the last non-missing value at or prior to the randomization. Change from BL was calculated by subtracting BL from the specific post-BL value. If BL or post-BL value was missing, the change from BL was set to missing.
Time Frame: Baseline and up to 36 weeks
Population: RD Full Analysis Population
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Randomized Placebo | Randomized Lamotrigine 200 mg/Day
Number analyzed (Participants) | 133 | 130
Score on a scale | 3.0 (0.83) | 1.8 (0.84)
Statistical Analysis 1: Comparison: Randomized Placebo vs Randomized Lamotrigine 200 mg/Day; Test type: Superiority or Other; p = 0.155, ANCOVA; Mean Difference (Final Values) = -1.2, 95% CI 2-sided [-3.0 to 0.5]

8. Secondary Outcome: Change From Baseline in Young Mania Rating Scale (YMRS) Total Score
Description: YMRS consists of 11 items: Elevated Mood, Increased Motor Activity/Energy, Sexual Interest, Sleep, Irritability, Speech, Language/Thought Disorder, Content, Disruptive/Aggressive Behaviour, Appearance, and Insight. Investigators rated par. from 0 to 4 (or 8) for each of these items. Total score is the sum of all subscales, from 0 to 60 (higher is worse). Data was collected on Wks 0, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 32, 36. Analysis was performed using ANCOVA with covariates of site, CGI-S BL score, treatment and YMRS total BL score. In LOCF datasets, the last non-missing OT score prior to TIME was carried forward to estimate missing data points for the remaining study visits of the treatment period. BL value was defined as the last non-missing values at or prior to the randomization. Change from BL at the time point of interest was calculated by subtracting BL value from the individual post-BL value. If either the BL or post-BL value was missing, change from BL was set to missing.
Time Frame: Baseline and up to 36 weeks
Population: RD Full Analysis Population
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Randomized Placebo | Randomized Lamotrigine 200 mg/Day
Number analyzed (Participants) | 133 | 130
Score on a scale | 2.4 (0.87) | 2.8 (0.88)
Statistical Analysis 1: Comparison: Randomized Placebo vs Randomized Lamotrigine 200 mg/Day; Test type: Superiority or Other; p = 0.661, ANCOVA; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-1.4 to 2.2]

9. Secondary Outcome: Change From Baseline of Global Assessment Scale (GAS) Total Score
Description: For GAS, investigators rated par. for lowest level of functioning during the previous week. The scale has a 10 score categories: 1-10, 11-20, 21-30, 31-40, 41-50, 51-60, 61-70, 71-80, 81-90, 91-100, using intermediary levels when appropriate (from 100 to 1, Lower is worse.). Data was collected on Weeks 0, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 32, 36. Analysis was performed using ANCOVA with covariates of site, CGI-S BL score, treatment and GAS total BL score. In presented LOCF datasets, the last non-missing on therapy score prior to TIME was carried forward to estimate missing data points for the remaining study visits of the treatment period. The BL value was defined as the last non-missing values at or prior to the randomization. The change from BL at the time point of interest was calculated by subtracting the BL values from the individual post-BL values. If either the BL or post-BL value was missing, the change from BL was set to missing as well.
Time Frame: Baseline and up to 36 weeks
Population: RD Full Analysis Population
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Randomized Placebo | Randomized Lamotrigine 200 mg/Day
Number analyzed (Participants) | 133 | 130
Score on a scale | -4.7 (1.75) | -4.9 (1.77)
Statistical Analysis 1: Comparison: Randomized Placebo vs Randomized Lamotrigine 200 mg/Day; Test type: Superiority or Other; p = 0.945, ANCOVA; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-3.7 to 3.5]

10. Secondary Outcome: Change From Baseline in Body Weight
Description: Participant's body weight was measured on Weeks 0, 4, 8, 12, 16, 20, 24, 32 and 36. Analysis was performed using ANCOVA with covariates of site, CGI-S baseline score, treatment and baseline body weight. In presented LOCF datasets, the last non-missing on therapy score prior to TIME was carried forward to estimate missing data points for the remaining study visits of the treatment period. The baseline value was defined as the last non-missing values at or prior to the randomization. The change from baseline at the time point of interest was calculated by subtracting the baseline values from the individual post-baseline values. If either the baseline or post-baseline value was missing, the change from baseline was set to missing as well.
Time Frame: Baseline and up to 36 weeks.
Population: RD Full Analysis Population. Only those par. with available data at indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Kilograms
Arm/Group | Randomized Placebo | Randomized Lamotrigine 200 mg/Day
Number analyzed (Participants) | 133 | 128
Kilograms | -0.72 (0.399) | -1.56 (0.407)
Statistical Analysis 1: Comparison: Randomized Placebo vs Randomized Lamotrigine 200 mg/Day; Test type: Superiority or Other; p = 0.047, ANCOVA; Mean Difference (Final Values) = -0.84, 95% CI 2-sided [-1.66 to -0.01]

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from the start of study treatment and until the follow up contact (up to Study Day 230).
Description: On-treatment SAEs and non-serious AEs were reported for the Safety population consisted of all participants who received at least one dose of study drug.
Arm/Group | Randomized Placebo | Randomized Lamotrigine 200 mg/Day
Serious Adverse Events (participants affected / at risk) | 3/133 | 2/131
Other Adverse Events (participants affected / at risk) | 46/133 | 40/131
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Randomized Placebo (N=133) | Randomized Lamotrigine 200 mg/Day (N=131)
Mania (Psychiatric disorders) | 2 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0
Brain stem infarction (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Randomized Placebo (N=133) | Randomized Lamotrigine 200 mg/Day (N=131)
Nasopharyngitis (Infections and infestations) | 4 | 4
Urinary tract infection (Infections and infestations) | 4 | 3
Upper respiratory tract infection (Infections and infestations) | 4 | 2
Herpes zoster (Infections and infestations) | 0 | 1
Pericoronitis (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Weight decreased (Investigations) | 1 | 3
Alanine aminotransferase increased (Investigations) | 2 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 2
Blood glucose increased (Investigations) | 2 | 1
Blood pressure increased (Investigations) | 2 | 1
Blood triglycerides increased (Investigations) | 2 | 0
Blood uric acid increased (Investigations) | 2 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 1
Weight increased (Investigations) | 2 | 0
Bilirubin conjugated increased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1
Blood phosphorus increased (Investigations) | 0 | 1
Blood urine present (Investigations) | 0 | 1
Electrocardiogram ST segment abnormal (Investigations) | 0 | 1
Electrocardiogram T wave abnormal (Investigations) | 1 | 0
Electrocardiogram abnormal (Investigations) | 0 | 1
Heart rate decreased (Investigations) | 0 | 1
Heart rate increased (Investigations) | 1 | 0
Neutrophil count increased (Investigations) | 1 | 0
Specific gravity urine increased (Investigations) | 0 | 1
Urine ketone body present (Investigations) | 0 | 1
White blood cell count increased (Investigations) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 2
Nausea (Gastrointestinal disorders) | 1 | 3
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Chronic gastritis (Gastrointestinal disorders) | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Lip ulceration (Gastrointestinal disorders) | 0 | 1
Retching (Gastrointestinal disorders) | 0 | 1
Headache (Nervous system disorders) | 4 | 4
Poor quality sleep (Nervous system disorders) | 4 | 2
Dizziness (Nervous system disorders) | 1 | 2
Somnolence (Nervous system disorders) | 1 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0
Depressed mood (Psychiatric disorders) | 2 | 1
Insomnia (Psychiatric disorders) | 2 | 1
Affect lability (Psychiatric disorders) | 1 | 0
Agitation (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Emotional distress (Psychiatric disorders) | 1 | 0
Hyposomnia (Psychiatric disorders) | 0 | 1
Initial insomnia (Psychiatric disorders) | 1 | 0
Irritability (Psychiatric disorders) | 1 | 0
Listless (Psychiatric disorders) | 1 | 0
Sleep disorder (Psychiatric disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 0
Fatigue (General disorders) | 3 | 2
Asthenia (General disorders) | 2 | 0
Chest discomfort (General disorders) | 0 | 1
Malaise (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Thirst (General disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 1
Bundle branch block right (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 1
Gout (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 2 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Granulocytopenia (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Dry eye (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 0
Thyroid disorder (Endocrine disorders) | 1 | 0
Food allergy (Immune system disorders) | 1 | 0
Menstrual disorder (Reproductive system and breast disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.